CLINICAL TRIAL: NCT05485402
Title: Foods Such as Virgin Olive Oil Rich in Phenolic Compounds, and Prebiotic Supplementation: Dietary Strategy to Tackle Sarcopenia in Early Elderly Subjects (FOOP-Sarc)
Brief Title: Dietary Strategy to Tackle Sarcopenia in Early Elderly Subjects (FOOP-Sarc)
Acronym: FOOP-Sarc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Rovira i Virgili (Other)
Responsible Party: Principal Investigator, Rosa Sola, Full Professor, Dr., University Rovira i Virgili
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FOOP-Sarc study; PID2019-105164RB-I00 (Other Grant/Funding Number: MCIN/AEI/10.13039/501100011033)
Record Dates: First submitted 2022-07-26; First posted 2022-08-03 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2023-05

CONDITIONS: Sarcopenia
Keywords: early elderly; olive oil; prebiotic supplementation; muscle mass; muscle strength; physical performance
MeSH Terms: conditions — Sarcopenia | interventions — 3,4-dihydroxyphenylethanol; maltodextrin; Prebiotics; Inulin

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, parallel and double-blind intervention study. The total duration of the study will be 24 weeks (12-weeks of intervention and 12-weeks of follow-up). The study will have three arms of intervention. The intervention products will be prebiotic supplement based on FOS and inulin or virgin olive oil rich in phenolic compounds with 156 mg hydroxytyrosol and tyrosol/kg oil. The placebo will be refined olive oil (38.6 mg hydroxytyrosol and tyrosol/kg oil) or maltodextrin. Both with the same format and appearance, to ensure the double-blind intervention.
  All the volunteers will receive NFOC-diet and physical activity recommendations co-created during the co-creation study. The nutritional recommendations are based on DASH diet and foods rich in protein (in particular, leucine), vitamin D, polyunsaturated acids, phosphorus and iron. The physical activity recommendations are 150 min/week of physical activity, with at least two sessions focused on motor strength.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Group A) (Placebo Comparator): Refined olive oil (38.6 mg hydroxytyrosol and tyrosol/kg oil), maltodextrin, and nutritional and physical activity recommendations
  Interventions: Dietary Supplement: Refined olive oil (38.6 mg hydroxytyrosol and tyrosol/kg oil); Dietary Supplement: Maltodextrin; Other: Nutritional and physical activity recommendations
- Intervention group (Group B) (Experimental): Virgin olive oil rich in phenolic compounds (156 mg hydroxytyrosol and tyrosol/kg oil), maltodextrin, and nutritional and physical activity recommendations
  Interventions: Dietary Supplement: Virgin olive oil rich in phenolic compounds (156 mg hydroxytyrosol and tyrosol/kg oil); Dietary Supplement: Maltodextrin; Other: Nutritional and physical activity recommendations
- Intervention group (Group C) (Experimental): Virgin olive oil rich in phenolic compounds (156 mg hydroxytyrosol and tyrosol/kg oil), prebiotic supplementation (FOS and inulin), and nutritional and physical activity recommendations
  Interventions: Dietary Supplement: Virgin olive oil rich in phenolic compounds (156 mg hydroxytyrosol and tyrosol/kg oil); Dietary Supplement: Prebiotic (FOS and inulin); Other: Nutritional and physical activity recommendations

INTERVENTIONS:
Dietary Supplement: Refined olive oil (38.6 mg hydroxytyrosol and tyrosol/kg oil) — The dosage will be 30 ml/day of refined olive oil (38.6 mg hydroxytyrosol and tyrosol/kg oil) used as a dressing (without heat).
  Arms: Control group (Group A)
Dietary Supplement: Virgin olive oil rich in phenolic compounds (156 mg hydroxytyrosol and tyrosol/kg oil) — The dosage will be 30 ml/day of virgin olive oil rich in phenolic compounds (156 mg hydroxytyrosol and tyrosol/kg oil) used as a dressing (without heat).
  Arms: Intervention group (Group B); Intervention group (Group C)
Dietary Supplement: Maltodextrin — The dosage will be 7,5 g/day of maltodextrin.
  Arms: Control group (Group A); Intervention group (Group B)
Dietary Supplement: Prebiotic (FOS and inulin) — The dosage will be 7,5 g/day of prebiotic supplement (FOS and inulin).
  Arms: Intervention group (Group C)
Other: Nutritional and physical activity recommendations — The nutritional recommendations are based on DASH diet and foods rich in protein (in particular, leucine) and vitamin D, polyunsaturated acids, phosphorus and iron. The physical activity recommendations are 150 min/week of physical activity, with at least two sessions dedicated to the development of motor strength.

SUMMARY:
The main objective of the present study is to add knowledge of the potential health effects and mechanism of action by a dietary strategy based on a VOO rich in phenolic compounds (156 mg hydroxytyrosol and tyrosol/kg oil) alone or combination with prebiotic supplementation based on fructooligosaccharides (FOS) and inulin to tackle sarcopenia by improving skeletal muscle mass and function and CVD risk factors in early elderly (60-80 years) home-dwelling sarcopenic subjects.

The specific objectives:

* To determine the compliance food intake biomarkers of VOO in 24h urine samples and prebiotic intake in faecal samples.
* To evaluate the effect of the NFOC-diet supplemented by VOO rich in phenolic compounds (156 mg hydroxytyrosol and tyrosol/kg oil) alone or in combination with prebiotic supplementation (FOS and inulin) on the improvement of muscle mass, muscle performance, gait performance, cardiovascular disease risk factors (inflammation, oxidation and endothelial function), and gut microbiota, in sarcopenic young-elderly subjects.
* To assess the mechanisms of action of the NFOC-diet supplemented by VOO rich in phenolic compounds (156 mg hydroxytyrosol and tyrosol/kg oil) alone or in combination with prebiotic supplementation (FOS and inulin) involved in the development of sarcopenia and cardiovascular disease in vivo and in vitro cellular models.
* To determine if the effects achieved after the intervention (12 weeks of intervention) will be sustained 12 weeks after the FOOP-Sarc intervention cessation (12 weeks of intervention + 12 weeks of follow-up), by assessing the sarcopenia and CVD risk factors in sarcopenic early elderly subjects.
* To co-create nutritional and physical activity recommendations of FOOP-Sarc study based on sarcopenia improvement by a sample of volunteers of the FOOP-Sarc study, and to assess the adherence and the effectivity of the recommendations, in comparison to standard recommendations created by researchers, the satisfaction and engagement experience in a co-creation process, and the usability of recommendations.

DETAILED DESCRIPTION:
The prebiotic supplementation about FOS and inulin was related to gut microbiota transformation an increase in handgrip strength and a reduction of exhaustion in older adults over 65 years old.

In the role of a nutritional intervention for the treatment of sarcopenia, an adequate intake of protein, especially leucine, vitamin D and antioxidant nutrients are recommended. In particular, dietary protein is a key anabolic stimulus for muscle protein synthesis. Moreover, food such as, virgin olive oil (VOO) can be involved in sarcopenia, by modulation of pro-inflammatory cytokines and could attenuate sarcopenic symptomology.

On the other hand, physical activity (PA) is an important aspect to avoid loss of muscle mass, for this reason, in sarcopenic subjects it is recommended to spend 150 min/week of moderate to vigorous physical activity.

A total of 39 home-dwelling early elderly volunteers will be included in the intervention (13 in each arm of the intervention). The total duration of the study will be 24 weeks (12-week period of dietary-lifestyle treatment and a 12-week period of follow-up after intervention cessation). Additionally, a total of 13 home-dwelling early elderly volunteers will be included in the co-creation process. Specifically, 7 home-dwelling early elderly volunteers will participate in the co-ideation and co-design steps. Additionally, 6 home-dwelling early elderly volunteers will participate in the co-implementation and comparison of recommendations (3 in each arm of intervention). The sample of volunteers that will co-implement will be randomized and different from the sample of volunteers that will co-ideate and co-design the recommendations. The co-evaluation step will include all 13 volunteers from the different steps of the co-creation process.

During the preliminary co-creation phase, there will be 5 visits over 6 weeks. A screening visit (V0) and one visit for each co-creation stage (co-ideation [V1], co-design [V2], co-implementation [V3] and co-evaluation [V4]). The volunteers who participated in the co-ideation and co-design stages had a total of 4 visits (V0, V1, V2 and the co-evaluation [V4] at the end of the co-design stage). The volunteers who participated in the co-implementation stage had a total of 3 visits (V0, V3 and V4).

Additionally, during the FOOP-Sarc study, there will be 6 visits in total (5 visits during the intervention period and 1 follow-up visit). Of these visits, 4 will be face-to-face and 3 by telephone. The study visits will be the following: screening visit (V0, face-to-face): to check inclusion/exclusion criteria and, in case of satisfying the inclusion criteria; basal visit (V1); visits during the intervention (V2, telephone; V3, telephone; V4, telephone); final study visit (V5, face-to-face); and follow-up visit (V6, face-to-face): follow-up visit 12-week after intervention cessation. In visits V0, V1, V5, and V6 volunteers must present themselves in fasting conditions of 8 hours to obtain blood. In visits V1, V5, and V6 volunteers must bring urine and feaces samples.

ELIGIBILITY:
Inclusion Criteria:

* Men and women with and age equal to or greater than 60 years and until 80 years.
* Written informed consent provided before the initial visit.
* Sarcopenia assessment: low muscle strength based on grip dynamometry, kg (men <30 kg; women <20 kg) or low skeletal muscle mass index (SMI) based on bioimpedance analysis (BIA), kg/m2 (men <8,87 kg/m2; women <6,42 kg/m2) or low physical performance or physical function based on 4m gait speed, m/s (≤0,8 m/s)

Exclusion Criteria:

* Type 2 or insulin-dependent diabetes diagnosed.
* Anemia (hemoglobin ≤13 g/dL in men and ≤12 g/dL in women).
* Intestinal malabsorption diseases.
* Fructose and/or sucrose intolerance.
* Malnutrition (assessed by albumin <3,5 g/dl).
* Renal diseases.
* Chronic alcoholism.
* Current or past participation in a clinical trial or consumption of a research product in the 30 days prior to inclusion in the study.
* Institutionalized elderly.
* Failure to follow the study guidelines.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Change in muscle mass | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  The change in muscle mass will be assess by the change in skeletal muscle mass index (kg/m2) measured by segmental multifrequency body composition analyser (TANITA MC-780MA; Tanita Corp., Tokyo, Japan)

SECONDARY OUTCOMES:
Body-weight | Visit 0 (week -1), visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Measured with calibrated scale in kg
Height | Visit 0 (week -1), visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Measured with wall-mounted stadiometer in cm
Body Mass Index | Visit 0 (week -1), visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Calculated by weight (kg) divided to height (m2)
Body weight composition | Visit 0 (week -1), visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Measured by segmental multifrequency body composition analyser (TANITA MC-780MA; Tanita Corp., Tokyo, Japan).
Waist circumference | Visit 0 (week -1), visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Steel measuring tape at the umbilicus in cm.
Sarcopenia assessment_skeletal muscle strength | Visit 0 (week -1), visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  grip strength, kg: Handheld dynamometer and the maximum value from either hand will be analyzed (Jamar dynamometer; Sammons Preston Rolyan, Bolingbrook, IL)
Sarcopenia assessment_muscle mass | Visit 0 (week -1), visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Muscle mass measured by segmental multifrequency body composition analyser (TANITA MC-780MA; Tanita Corp., Tokyo, Japan)
Sarcopenia assessment_muscle physical performance | Visit 0 (week -1), visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Gait speed, m/s: length of the walking course divided by the time
Compliance of physical activity recommendations | Visit 1 (week 0), visit 2 (week 3), visit 3 (week 6), visit 4 (week 9) visit 5 (week 12), visit 6 (week 24)
  IPAQ-E Spanish version
Compliance of the dietary recommendations | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Dietary record: 3-day dietary record
Dietary compliance markers | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Folin-Ciocalteau method adjusted by creatinine values, measured in 24h urine samples
Specific phenolic compounds_dietary compliance markers | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Specific phenolic compounds and metabolites assessed by Ultra performance liquid chromatography - tandem mass spectrometer (UPLC-MS/MS) in urine samples
Phenolic metabolites_dietary compliance markers | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Phenolic metabolites by UPLC-MS/MS in plasma
Sarcopenia and Quality of life | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  SarQoL® test assessed by quality of life test adapted to sarcopenic subjects. It is scored from 0 to 100, where higher values indicate better quality of life.
Fasting blood glucose (FBG) | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  by standardized methods in an automated analyzer (Beckman Coulter-Synchron, Galway, Ireland) in (mmol/L)
Insulin | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  by standardized methods in an automated analyzer (Beckman Coulter-Synchron, Galway, Ireland) in (IU/mL)
Homeostasis model assessment index (HOMA index) | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Calculated by fasting insulin (μUI/mL) x fasting glucose (mmol/L) / 22,5
Lipid profile | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Total cholesterol (TC), high density lipoprotein cholesterol (HDLc), low density lipoprotein cholesterol (LDLc) and Total triglycerides (TG) in mmol/L by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Apolipoproteins | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Apolipoprotein A1 (ApoA1) and apolipoprotein B100 (ApoB100) in mg/dL by standardized enzymatic automated methods in an autoanalyzer (Beckman Coulter-Synchron, Galway, Ireland)
Apolipoproteins ratio | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Calculated by ApoA1 divided to ApoB100
Vascular parameters_endothelial function | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Ischemic reactive hyperemia (IRH) with Laser-Doppler Linear Periflux 5000 (Perimed AB, Järfälla, Stockholm, Sweden)
Vascular parameters_blood pressure | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Systolic blood pressure (SBP) and Diastolic blood pressure (DBP) in mm Hg by automatic sphygmomanometer (OMRON HEM-907; Peroxfarma, Barcelona, Spain).
Vascular parameters_pulse pressure | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Calculated by SBP - DBP
Endothelin | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Endothelin in pg/mL assessed by Commercial ELISA
Endothelial dysfunction markers | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  E-selectin (CD62E), P-selectin (CD62P), Intercellular Cell Adhesion Molecule 1 (ICAM-1 (CD54)) and Vascular Cell Adhesion Molecule 1 (VCAM-1 (CD106) assessed by multi-analyte ELISArray kits.
Oxidative biomarkers_Oxidized LDL | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Oxidized LDL (oxLDL) assessed by commercial ELISA.
Oxidative biomarkers_Superoxide Dismutase | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Superoxide Dismutase (SOD) in U/g Hb assessed by enzymatic assay
Oxidative biomarkers_Glutathione peroxidase | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Glutathione peroxidase (GSHPx) in nmol/mL assessed by enzymatic assay
Inflammation biomarkers_High sensitivity C-reactive protein | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  High sensitivity C-reactive protein (hsCRP) in mg/L assessed by Immunoturbidimetry on an autoanalyzer (Roche Diagnostics Systems, Madrid, Spain)
Inflammation biomarkers_interleukine-6 | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Interleukine-6 (IL-6) in pg/mL assessed by Immunoturbidimetry on an autoanalyzer (Roche Diagnostics Systems, Madrid, Spain)
Inflammation biomarkers_uric acid | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Uric acid in mg/dL is assessed by Immunoturbidimetry on an autoanalyzer (Roche Diagnostics Systems, Madrid, Spain)
Inflammation biomarkers_tumour necrosis factor-α | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Tumour necrosis factor-α (TNF-α) in pg/mL is assessed by commercial ELISA kit.
Renal function_creatinine | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Creatinine in mg/dL is assessed by standardized methods in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain) in 24 h urine samples
Renal function_glomerular filtration rate | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Glomerular filtration rate (GFR) in mL/minutes/1.73m2 is assessed by equation Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI).
Endocrine system | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Testosterone (pg/mL) and growth hormone (GH) (pg/mL)) assessed by in a Cobas Mira Plus autoanalyzer (Roche Diagnostics Systems, Madrid, Spain)
Proteome profiling | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Whole proteome assessed by nano Liquid chromatography-mass spectrometry (nLC-MS) according to our previous work.
Gut microbiota_phyla composition and functionality | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Phyla composition and functionality assessed by whole genomic content sequencing. Illumina platform will be used to obtain the metagenomics and metatranscriptomics of each sample following previous protocols developed in Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (FISABIO-Salud Pública (Valencia)).
Gut microbiota_short chain fatty acids | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Short chain fatty acids (SCFA): bile acids, sterols, buthyrate, and branched chain amino acids and sterols assessed by gas chromatography (GC)
wasting and turnover | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Myostatin, follistatin, and ratio myostatin/follistatin in serum samples will be measured at V1 and V5 by Human Myostatin MSTN ELISA Kit and Human Follistatin Like Protein 1 (FSTL1) ELISA Kit.
Muscle mass ultrasound assessment | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Muscle mass assessment will be assessed based on dominant upper leg ultrasound. The measurements will be: Subcutaneous adipose tissue thickness (cm); quadriceps muscle thickness (cm); rectus femoris muscle thickness (Y axis) (cm) and cross-sectional area (cm2); pennation angle (º).
  Ultrasound assessment will be conducted by VINNO 5 (Vinno (Suzhou) Co., Ltd., China) at HAR-mode with the musculoskeletal (MSK) superficial preset at a frequency of 10 MHz with a linear transducer (Vinno (Suzhou) Co., Ltd., China).
Muscle mass isokinetic assessment | Visit 1 (week 0), visit 5 (week 12)
  Muscle mass assessment will be carried out with an isokinetic dynamometer (Biodex System 4; Biodex Medical Systems, New York, USA) based on dominant upper leg.
  The parameters assessed at an angular velocity of 180º s-1 and 240º s-1 in leg extension and flexion will be: maximum peak torque (N m), maximum total work (J), mean power (W) and the ratio between the mean power by isokinetic and the rectus femoris cross-sectional area by ultrasound.
Frailty | Visit 1 (week 0), visit 5 (week 12), visit 6 (week 24)
  Frailty will be assessed by Fried criteria

CONTACTS AND LOCATIONS:
Overall Officials: Rosa Solà, Dr, Principal Investigator — University Rovira i Virgili, Reus, Tarragona, Spain; Rosa Maria Valls, Dr, Principal Investigator — University Rovira i Virgili, Reus, Tarragona, Spain
Locations (1):
- Universitat Rovira i Virgili, Reus, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubio Castaneda FJ, Tomas Aznar C, Muro Baquero C. [Validity, Reliability and Associated Factors of the International Physical Activity Questionnaire Adapted to Elderly (IPAQ-E)]. Rev Esp Salud Publica. 2017 Jan 18;91:e201701004. Spanish. PMID 28098134
- [Background] Ignacio de Ulibarri J, Gonzalez-Madrono A, de Villar NG, Gonzalez P, Gonzalez B, Mancha A, Rodriguez F, Fernandez G. CONUT: a tool for controlling nutritional status. First validation in a hospital population. Nutr Hosp. 2005 Jan-Feb;20(1):38-45. PMID 15762418
- [Background] Beaudart C, Biver E, Reginster JY, Rizzoli R, Rolland Y, Bautmans I, Petermans J, Gillain S, Buckinx F, Dardenne N, Bruyere O. Validation of the SarQoL(R), a specific health-related quality of life questionnaire for Sarcopenia. J Cachexia Sarcopenia Muscle. 2017 Apr;8(2):238-244. doi: 10.1002/jcsm.12149. Epub 2016 Oct 22. PMID 27897430
- [Background] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jan 1;48(1):16-31. doi: 10.1093/ageing/afy169. PMID 30312372
- [Derived] Besora-Moreno M, Sepulveda C, Queral J, Jimenez-Ten Hoevel C, Pedret A, Tarro L, Valls RM, Sola R, Llaurado E. Participatory Research in Clinical Studies: An Innovative Approach to Co-creating Nutritional and Physical Activity Recommendations for Older Adults With Sarcopenia (FOOP-Sarc Project). Health Expect. 2025 Apr;28(2):e70187. doi: 10.1111/hex.70187. PMID 40184328
- [Derived] Besora-Moreno M, Llaurado E, Jimenez-Ten Hoevel C, Sepulveda C, Queral J, Bernal G, Perez-Merino L, Martinez-Hervas S, Alabadi B, Ortega Y, Valls RM, Sola R, Pedret A. New Perspectives for Low Muscle Mass Quantity/Quality Assessment in Probable Sarcopenic Older Adults: An Exploratory Analysis Study. Nutrients. 2024 May 15;16(10):1496. doi: 10.3390/nu16101496. PMID 38794734